CLINICAL TRIAL: NCT00367809
Title: Impact of Mind-Body Interventions Post Organ Transplant
Brief Title: Wellness Interventions After Transplant Study
Acronym: WIAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Cynthia R. Gross, Professor, University of Minnesota, College of Pharmacy and School of Nursing
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GCRC Protocol 942
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Organ Transplant
Keywords: Meditation; Mindfulness; Organ Transplant; Transplantation; Minnesota; Immune suppressive therapy
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MSBR)
- 2 (Active Comparator)
  Interventions: Behavioral: Health Education (HE)
- 3 (No Intervention)
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MSBR) — Mindfulness-Based Stress Reduction (MBSR) is the intervention of primary interest. It is a psycho-educational program of 8-weekly classes, 2.5 hours long taught by a trained instructor. Over the course of the program participants receive training in several formal meditation techniques: a body-scan meditation, sitting meditation, walking meditation and mindful Hatha yoga that involves simple stretches and movements. Participants are requested to practice meditation at home and to integrate informal mindfulness practices into their daily lives. The content of MBSR is described in the book Full Catastrophe Living by Jon Kabat-Zinn.
  Arms: 1
Behavioral: Health Education (HE) — The active control condition was a peer-led chronic disease self-management program comprised of 8 weekly, 2.5 hour meetings. Led by trained peer-leaders, groups of participants discussed health challenges and problem-solved using a technique called action-planning. The curriculum described by Lorig and colleagues in the book Living a Health Life was the core of this program, and transplant-specific issues were covered in two meetings to match MBSR for time and attention.
  Arms: 2
Behavioral: Delayed Intervention — A temporary wait-list control group; after 6 months, those in the Delayed Intervention were randomized a second time, to one of the active treatment arms (MBSR or HE).
  Arms: 3

SUMMARY:
The Wellness Interventions after Transplant (WIAT) Trial has reached its enrollment target. This trial is no longer recruiting new patients. Those currently enrolled will be followed for a year to evaluate trial outcomes.

The purpose of this trial is to determine if training in Mindfulness-Based Stress Reduction can reduce symptom distress and improve quality of life in solid organ transplant recipients. Primary study outcomes are depression, anxiety and insomnia symptoms, measured by well-validated self-report scales. The impact of this program on objectively measured sleep outcomes, use of health care resources and costs will also be evaluated.

DETAILED DESCRIPTION:
Pharmacologic options for managing symptoms increase the risks of side effects and drug interactions, and may reduce adherence by complicating an already challenging medication regimen. In contrast, mind-body based complementary therapies may be ideal to treat distressing symptoms and negative emotions after transplantation. Our long-range objective is to develop evidence-based recommendations for non-pharmacologic strategies that provide symptom relief to transplant recipients, and are safe, practical and cost-effective.

Potential participants are recruited by mail, screening by clinic staff and provider referrals. Interested persons are screened by telephone and mailed informational study brochures. Informed consent is conducted by face-to-face interview, where a diagram of the study design is used to explain the 2-stage randomization and study requirements.

ELIGIBILITY:
Inclusion Criteria:

* kidney, kidney/pancreas, pancreas, lung, liver, heart or heart-lung recipients, with a functioning graft
* 18 years old or older
* English-speaking
* literate
* mentally intact
* reachable by telephone
* on immune suppressive medication
* receiving regular medical follow-up care
* interested in health promotion and mind-body interventions
* able to attend weekly classes in a Minnesota Metro area
* willing to complete the informed consent process

Exclusion Criteria:

* serious preexisting mental health issues such as suicide attempts or a psychosis
* medically unstable (a hospital admission for non-elective purposes in the last 3 months or major surgery planned in the next 3 months)
* on dialysis
* regularly practicing mindfulness meditation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduction in depression | Baseline; at 8 weeks, at 6- and 12- months
anxiety | Baseline; at 8 weeks, at 6- and 12- months
insomnia | Baseline; at 8 weeks, at 6- and 12- months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Cynthia Gross, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Academic Health Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Gross CR, Kreitzer MJ, Russas V, Treesak C, Frazier PA, Hertz MI. Mindfulness meditation to reduce symptoms after organ transplant: a pilot study. Altern Ther Health Med. 2004 May-Jun;10(3):58-66. PMID 15154154
- [Result] Kreitzer MJ, Gross CR, Ye X, Russas V, Treesak C. Longitudinal impact of mindfulness meditation on illness burden in solid-organ transplant recipients. Prog Transplant. 2005 Jun;15(2):166-72. doi: 10.1177/152692480501500210. PMID 16013466
- [Derived] Gross CR, Kreitzer MJ, Thomas W, Reilly-Spong M, Cramer-Bornemann M, Nyman JA, Frazier P, Ibrahim HN. Mindfulness-based stress reduction for solid organ transplant recipients: a randomized controlled trial. Altern Ther Health Med. 2010 Sep-Oct;16(5):30-8. PMID 20882729
- [Derived] Gross CR, Kreitzer MJ, Reilly-Spong M, Winbush NY, Schomaker EK, Thomas W. Mindfulness meditation training to reduce symptom distress in transplant patients: rationale, design, and experience with a recycled waitlist. Clin Trials. 2009 Feb;6(1):76-89. doi: 10.1177/1740774508100982. PMID 19254938